CLINICAL TRIAL: NCT05469360
Title: A Randomized, Participant and Investigator Blinded, Placebo-Controlled Study to Evaluate the Ability of a Single Intrathecally Administered Dose of NIO752 to Lower Cerebrospinal Fluid Total Tau Levels in Participants With Early Alzheimer's Disease
Brief Title: Study of Safety, Tolerability, Pharmacodynamics and Pharmacokinetics of NIO752 in Early Alzheimer's Disease Participants
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: CNIO752B12201; 2024-514004-14 (Other: EU CTIS)
Record Dates: First submitted 2022-07-11; First posted 2022-07-21 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2025-08

CONDITIONS: Alzheimer Disease; Mild Cognitive Impairment
Keywords: Alzheimer Disease; Autosomal dominant Alzheimer disease; Early onset Alzheimer disease; Familial Alzheimer disease; Dementia; Brain Diseases; Central Nervous System Diseases; Nervous System Diseases; Tauopathies; Neurodegenerative Diseases; Neurocognitive Disorders; Memory loss; Placebo; Adult
MeSH Terms: conditions — Alzheimer Disease; Cognitive Dysfunction; Dementia; Brain Diseases; Central Nervous System Diseases; Nervous System Diseases; Tauopathies; Neurodegenerative Diseases; Neurocognitive Disorders; Memory Disorders

STUDY DESIGN:
Intervention Model Description: Phase 1b
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- NIO752 - Dose A - Cohort 1 (Experimental): A single intrathecal injection of Dose A
  Interventions: Drug: NIO752
- Matching placebo - Cohort 1 (Placebo Comparator): A single intrathecal injection of artificial cerebrospinal fluid (CSF)
  Interventions: Drug: Matching placebo
- NIO752 Dose B - Cohort 2 (Experimental): A single intrathecal injection of Dose B
  Interventions: Drug: NIO752
- Matching placebo - Cohort 2 (Placebo Comparator): A single intrathecal injection of artificial cerebrospinal fluid (CSF)
  Interventions: Drug: Matching placebo
- NIO752 OLE - Cohorts 1 and 2 (Experimental): Multiple intrathecal injections of Dose A
  Interventions: Drug: NIO752
- NIO752 - Dose C - Cohort 3 (Experimental): Two intrathecal injections of Dose C
  Interventions: Drug: NIO752
- Matching Placebo - Cohort 3 (Placebo Comparator): Two intrathecal injections of artificial cerebrospinal fluid (CSF)
  Interventions: Drug: Matching placebo
- NIO752 OLE - Cohort 3 (Experimental): Single intrathecal injection of Dose C
  Interventions: Drug: NIO752

INTERVENTIONS:
Drug: NIO752 — A single intrathecal (cerebrospinal) injection of NIO752 of Dose A
  Arms: NIO752 - Dose A - Cohort 1
Drug: NIO752 — A single intrathecal (cerebrospinal) injection of NIO752 at dose B
  Arms: NIO752 Dose B - Cohort 2
Drug: Matching placebo — A single intrathecal injection of matching placebo
  Arms: Matching placebo - Cohort 1; Matching placebo - Cohort 2
Drug: NIO752 — Multiple intrathecal injections of NIO752 of Dose A
  Arms: NIO752 OLE - Cohorts 1 and 2
Drug: NIO752 — Two intrathecal injections of NIO752 at dose C
  Arms: NIO752 - Dose C - Cohort 3
Drug: NIO752 — Single intrathecal injection of NIO752 at dose C
  Arms: NIO752 OLE - Cohort 3
Drug: Matching placebo — Two intrathecal injections of matching placebo
  Arms: Matching Placebo - Cohort 3

SUMMARY:
Phase 1b study to assess the pharmacodynamics, safety, tolerability, and pharmacokinetics of NIO752 in patients with early Alzheimer's disease (AD)

DETAILED DESCRIPTION:
This is a phase 1b, randomized, double-blind, placebo-controlled study, in which 36 patients with early AD will be enrolled in one of three cohorts.

Cohorts 1 & 2 will receive a single intrathecal (IT) dose of NIO752 or placebo in the placebo-controlled part of the study, and multiple administrations of NIO752 in the open-label extension (OLE) part of the study.

Cohort 3 will receive two single IT doses of NIO752 or placebo in the placebo-controlled part of the study, and a single administration of NIO752 in the OLE part of the study.

Each cohort will enroll 12 participants, and they will be randomized into receiving NIO752 or placebo in 2:1 ratio. Participants in cohorts 1& 2 will remain in this study for approximately ~19 months, including ~18 in-clinic follow up visits during that period of time. In cohort 3, participants will remain in this study for a follow up period of approximately ~18 months including ~10 in-clinic follow up visits.

Cohorts will be enrolled sequentially.

Participants who complete the placebo-controlled part of the study will be eligible to continue in an OLE part of the study regardless of randomization assignment in the placebo-controlled part. All OLE participants will receive either two (cohorts 1 & 2) or one (cohort 3) dose of NIO752.

Study assessments will include physical and neurological examinations, ECGs, vital signs, standard clinical laboratory evaluations (hematology, blood chemistry, and urinalysis), routine laboratory evaluation of CSF collected through lumbar puncture, adverse event, and serious adverse event monitoring. Cohort 3 participation will also require 3 MRI scans and 3 PET scans throughout the 18 months of the study.

ELIGIBILITY:
Main Inclusion Criteria (placebo-controlled part):

* Between 30 to 74 years old (both inclusive) at the time of informed consent.
* A diagnosis of mild Alzheimer's Disease (AD) or mild cognitive impairment (MCI) due to AD at screening with at least a 6-month decline in cognitive function prior to screening documented in the medical record. Both participants with sporadic AD as well as Amyloid Precursor Protein (APP), Presenilin-1 (PSEN1) or Presenilin-2 (PSEN2) mutation carriers are eligible.
* Participants must have a diagnosis of MCI due to AD or mild AD at screening as defined by a Clinical Dementia Rating Scale (CDR) Global Score of 0.5 or 1 and a Memory Score ≥ 0.5.
* A history of CSF biomarkers supporting the diagnosis of AD obtained at any time point prior to screening, including CSF amyloid (amyloid-β 42 and/or 42/40 ratio) AND tau species (total tau and/or phosphorylated tau). All participants must have documented historical confirmation of both CSF biomarkers (amyloid-β and tau species) with results supporting a diagnosis of AD prior to screening. This criterion will be determined individually for each participant taking into consideration the biomarker assay used in each case. For participants (Cohorts 1 & 2 only) with no historical CSF biomarker information, a LP for CSF collection must be performed at the screening visit. For CSF collected at screening, participants must have confirmed positivity of amyloid-β-42 ≤ 1000 pg/mL as well as positivity on, at least, one of the following Tau biomarkers: phosphorylated-tau-181 > 12 pg/ml OR T-tau > 149.9 pg/mL as determined by the central laboratory.
* Participant has a reliable study partner or caregiver (e.g., spouse, sibling, close friend, adult child) who, is at least 18 years old.
* Participant resides in a proximity to the study site to allow a timely unscheduled visit to the study site, if necessary.
* Participant is able to undergo lumbar puncture (LP), CSF collections, and blood draws, tolerate brain MRI and PET scanning, and able to participate and tolerate all study procedures at study visit.

Main Inclusion Criteria (OLE part):

* Signed informed consent of protocol version inclusive of the OLE.
* Participant must complete Day 170 of the placebo-controlled part of this study.

Main Exclusion Criteria (placebo-controlled part):

* Participant lives in a skilled nursing facility or dementia care facility.
* Any previous use of experimental therapy within 180 days or 5 half-lives prior to Day 1, whichever is greater. Previous exposure to anti-tau and anti-β-amyloid antibodies is allowed if at the time of screening at least 180 days have passed since the last dose. Previous exposure to amyloid vaccines or tau vaccines meant to treat AD, or previous treatment with oligonucleotides or with gene therapy at any time frame is not allowed.
* Any current or past non-AD neurological conditions.
* Other medical conditions including but not limited to poorly controlled diabetes mellitus, unstable angina, myocardial infarction, chronic heart failure, clinical significant conduction abnormalities, impaired renal or kidney function, which, in the opinion of the Investigator, would make the participant unsuitable for inclusion or could interfere with the participation in or completion of the study.
* Treatment with immunosuppressants, antipsychotics, lithium, neuroleptics, dopaminergic agonists, L-dopa, or monoamine oxidase inhibitors at the time of screening. Current use of medications, other than cholinesterase inhibitors and/or memantine, that could alter cognition, as determined by the Investigator. If the participant is receiving cholinesterase inhibitors and/or memantine, the dose must have been stable within 12 weeks prior to screening, and must remain stable during the duration of the study.
* Brain MRI at screening or within 12 months prior to screening showing evidence of cerebrovascular disease such as acute or sub-acute micro- or macrohemorrhage, significant signs of major cerebrovascular disease, or any other imaging evidence that, in the opinion of the Investigator, makes the participant unsuitable for the study.

Main Exclusion Criteria (OLE part):

* Use of any investigational drugs, or participation in a clinical trial with an investigational new drug (other than NIO752), after completing the initial placebo-controlled part of this trial
* Participants who withdrew informed consent while participating in the main placebo-controlled part of the study

Ages: 30 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2023-02-23 (Actual); Primary Completion 2026-09-11 (Estimated); Study Completion 2028-01-02 (Estimated)

PRIMARY OUTCOMES:
Change in cerebrospinal total tau from baseline to Day 85 | Baseline, Day 85
  Total tau protein levels in cerebrospinal fluid. More frequent timepoints might be added as deemed necessary per the site Investigator's judgment.

SECONDARY OUTCOMES:
Number of adverse events and serious adverse events | Cohort 1 & 2: Baseline up to 170 days (placebo-controlled part) and up to 589 days (OLE part), Cohort 3: Baseline up to 169 days (placebo-controlled part) and up to 507 days (OLE part)
  Adverse events are assessed at each clinic visit. Laboratory values and other safety assessment values considered clinically significant by the investigator and meet the definition of adverse event will be reported.
Concentration of NIO752 in cerebrospinal fluid (CSF) | Cohorts 1 & 2: Pre-dose, Days 57, 85, 170 (placebo-controlled part) and Days 252, 420, and 588 (OLE part), Cohort 3: Pre-dose, day 1, 57, 85, 169 (placebo-controlled part) and Days 388 and 506 (OLE part)
  Concentration of NIO752 in CSF
Cmax, Ctrough in plasma | Cohorts 1, 2 & 3: Pre-dose, 0.5, 1, 2, 3 4, 5, 6, 24 hours post first dose. Cohort 1 & 2: Days 14, 57, 85 and 170 (pbo-controlled part) and 252, 253, 420, 421, and 588 (OLE) Cohort 3: Days 14, 57, 85 and 169 (pbo-controlled part) and 338 and 506 (OLE)
  Maximum and trough level concentrations of NIO752 in plasma
Tmax in blood plasma | Cohorts 1, 2 & 3: Pre-dose, 0.5, 1, 2, 3 4, 5, 6, 24 hours post first dose. Cohort 1 & 2: Days 14, 57, 85 and 170 (pbo-controlled part) and 252, 253, 420, 421, and 588 (OLE) Cohort 3: Days 14, 57, 85 and 169 (pbo-controlled part) and 338 and 506 (OLE)
  Time of Cmax in plasma post-IT injection
AUC-last in blood plasma | Cohorts 1, 2 & 3: Pre-dose, 0.5, 1, 2, 3 4, 5, 6, 24 hours post first dose. Cohort 1 & 2: Days 14, 57, 85 and 170 (pbo-controlled part) and 252, 253, 420, 421, and 588 (OLE) Cohort 3: Days 14, 57, 85 and 169 (pbo-controlled part) and 338 and 506 (OLE)
  Area under curve (AUC) from time zero to the last measurable concentration sampling time (t-last) (mass x time x volume-1)
AUC-inf in blood plasma | Cohorts 1, 2 & 3: Pre-dose, 0.5, 1, 2, 3 4, 5, 6, 24 hours post first dose. Cohort 1 & 2: Days 14, 57, 85 and 170 (pbo-controlled part) and 252, 253, 420, 421, and 588 (OLE) Cohort 3: Days 14, 57, 85 and 169 (pbo-controlled part) and 338 and 506 (OLE)
  The AUC from time zero to infinity (mass x time x volume-1)
Change in CSF total Tau | Cohorts 1 & 2: Pre-dose, Days 57, 85, 170 (placebo-controlled part) and Days 252, 420, and 588 (OLE part), Cohort 3: Pre-dose, day 1, 57, 85, 169 (placebo-controlled part) and Days 388 and 506 (OLE part)
  Evaluating the ability of NIO752 to lower CSF total tau in participants with early AD when administered as multiple doses

CONTACTS AND LOCATIONS:
Overall Officials: Madhav Thambisetty, MD PhD, Study Director — Novartis Pharmaceuticals
Locations (9):
- Finland (2):
  - Novartis Investigative Site, Kuopio
  - Novartis Investigative Site, Turku
- France (3):
  - Novartis Investigative Site, Lille
  - Novartis Investigative Site, Paris
  - Novartis Investigative Site, Toulouse
- Spain (2):
  - Novartis Investigative Site, Valencia, Valencia
  - Novartis Investigative Site, Barcelona
- Sweden (2):
  - Novartis Investigative Site, Malmo
  - Novartis Investigative Site, Stockholm

IPD SHARING:
Plan to Share IPD: No